CLINICAL TRIAL: NCT06170489
Title: A Phase III, Randomised, Open-label,, Multi-Center Clinical Study Comparing JS004 Plus Toripalimab With Investigator-Selected Chemotherapy in Patients With PD-(L)1 Monoclonal Antibody Refractory Classic Hodgkin Lymphoma (cHL)
Brief Title: A Phase III Clinical Study Comparing JS004 Plus Toripalimab With Investigator-Selected Chemotherapy in Patients With PD-(L)1monoclonal Antibody Refractory Classic Hodgkin Lymphoma (cHL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS004-009-III-cHL
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — toripalimab; Bendamustine Hydrochloride; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS004 plus Toripalimab (Experimental): JS004 200mg plus Toripalimab 240mg IV on day 1 of each cycle, every 3 weeks for up to 2 years
  Interventions: Biological: JS004 in combination with Toripalimab
- Investigator-Selected Chemotherapy (Active Comparator): Bendamustine or gemcitabine
  Interventions: Drug: Bendamustine or gemcitabine

INTERVENTIONS:
Biological: JS004 in combination with Toripalimab — Participants will receive JS004 in combination with Toripalimab (200 mg/240 mg) by intravenous (IV) infusion on Day 1, then every three weeks (Q3W), for up to 35 infusions.
  Arms: JS004 plus Toripalimab
Drug: Bendamustine or gemcitabine — Participants will receive Investigator-Selected chemotherapy of EITHER bendamustine by IV infusion at a dose of 90 or 120 mg/m^2 on Day 1 and Day 2 of either a 3- or 4-week cycle for up to 6 cycles OR gemcitabine by IV infusion at a dose of 1000 mg/m^2 on Day 1 and Day 8 of a 3-week cycle for up to 6 cycles.
  Arms: Investigator-Selected Chemotherapy

SUMMARY:
The study is being conducted to compare JS004 plus Toripalimab with Investigator-Selected Chemotherapy in Patients with PD-(L)1 monoclonal antibody refractory Classic Hodgkin Lymphoma (cHL)

DETAILED DESCRIPTION:
The study is a randomized, open-label, phase III clinical trial. The main objective is to compare the efficacy of JS004 plus Toripalimab with Investigator-Selected Chemotherapy in treating patients with PD-(L)1 monoclonal antibody refractory Classic Hodgkin Lymphoma (cHL). The study will assess the safety and tolerability of JS004 combined with Toripalimab.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled:

* Age at least 18 years old, both males and females are eligible
* Pathologically confirmed classical Hodgkin Lymphoma (cHL) with either relapsed (disease progression after achieving CR/PR in recent treatment) or refractory (failure to achieve CR/PR in recent treatment) status.
* Has exhausted all standard treatment and refractory to PD-(L)1 monoclonal antibody (mAb)
* ECOG: 0-2
* At least one measurable lesion meeting the criteria specified in the Lugano 2014 response assessment.

Exclusion Criteria:

* Known allergy or contraindication to the investigational drug or its components
* Permanent discontinuation of anti-PD-(L)1 antibody due to immune-related adverse reactions.
* Presence of central nervous system (CNS) metastasis.
* Presence of pleural effusion, ascites, or pericardial effusion requiring intervention (e.g., aspiration, drainage)
* Active autoimmune diseases requiring systemic treatment (such as corticosteroids or immunosuppressive drugs) within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per Lugano criteria 2014 as Assessed by Independent review committee (IRC) | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per Lugano criteria 2014 as assessed by IRC or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 45 months
  OS is defined as the time from randomization to death due to any cause.
Progression Free Survival (PFS) per Lugano criteria 2014 Assessed by Investigator | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per Lugano criteria 2014 assessed by Investigator or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) per Lugano criteria 2014 Assessed by Investigator | Up to approximately 36 months
  ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano criteria 2014 assessed by Investigator
Complete response rate (CRR) per Lugano criteria 2014 Assessed by Investigator | Up to approximately 36 months
  Complete response rate (CRR) is defined as the proportion of subjects in which BoR is CR, best overall response (BoR) refers to the best response as determined by the investigator.
Duration of Response (DOR) per Lugano Response Criteria as Assessed by Investigator | Up to approximately 36 months
  For participants who demonstrate CR or PR per Lugano criteria 2014 as assessed by Investigator, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Incidence and severity of all adverse events (AE) that occurred during the clinical trial | Up to approximately 36 months
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number and sverity of participants who experience an AE will be presented.
PK | Up to approximately 36 months
  To characterize the trough concentrations of JS004 and toripalimab;
Immunogenicity profiles | Up to approximately 36 months
  To characterize incidence and titer of antidrug antibodies (ADA) and/or neutralizing antibodies (Nab);

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No